CLINICAL TRIAL: NCT07282002
Title: Feasibility Protocol for Percutaneous AngioVac Vegetation Extraction (PAVE) to Remove Right Heart Vegetations in Patients With Infective Endocarditis
Brief Title: Percutaneous AngioVac Vegetation Extraction (PAVE) to Remove Right Heart Vegetations in Patients With Infective Endocarditis
Acronym: PAVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-CAR-01
Record Dates: First submitted 2025-11-20; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Infective Endocarditis (IE)
Keywords: AngioVac; Infective endocarditis (IE)
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AngioVac System (Experimental): Percutaneous removal of right-heart vegetation using the AngioVac System Cannula and Circuit
  Interventions: Device: AngioVac System

INTERVENTIONS:
Device: AngioVac System — Percutaneous vacuum-assisted aspiration of right-sided vegetation via suction, filtration and veno-venous bypass.

SUMMARY:
The investigation aims to demonstrate initial safety and efficacy of the AngioVac System for the removal of vegetation in the right heart in patients with infective endocarditis.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm investigational device study evaluating safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥ 18 years
2. Subject provides a signed and dated Informed Consent Form
3. Subject has a diagnosis of native infective endocarditis
4. Subject has presence of bacteremia with valvular (tricuspid or pulmonic) vegetations > 1 cm confirmed by transesophageal echocardiogram (TEE) or transthoracic echocardiogram (TTE) with the presence of septic emboli
5. Subject has no underlying terminal illness and subject is deemed medically eligible for interventional procedure(s) per institutional guidelines and/or clinical judgment

Exclusion Criteria:

1. Subject requires debulking of vegetation on cardiac leads
2. Subject has a prior history of ischemic/hemorrhagic stroke (within 3 months)
3. Subject has a coagulation disorder
4. Subject has arterial septic emboli
5. Subject has cerebral septic embolism
6. Subject has preoperative intubation due to ongoing hypoxemic respiratory failure
7. Subject has fungal endocarditis
8. Subject has atrial septal defect
9. Subject has medically refractory right-sided heart failure secondary to valvular dysfunction (SCAI SHOCK Stage Classification D or E)
10. Subject has planned valvular replacement/repair
11. Subject has prosthetic valves and/or annular abscesses
12. Subject has epidural abscesses
13. Subject is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Rate of Clinical Success | 30 days post-procedure
  The number and proportion of patients who experience clinical success, defined as a composite of 30-day survival, absence of persistent bacteremia within 30 days post-procedure, and absence of further right-sided valve intervention through 30 days post-procedure
Rate of Major Adverse Events (MAEs) | 48 hours post-procedure
  The number and proportion of subjects who experience a MAE within 48 hours post-procedure. MAEs include: all-cause mortality, major bleeding, and device- or procedure-related adverse events of cardiac perforation, vascular perforation, dissection, or pericardial effusion/tamponade

SECONDARY OUTCOMES:
Proportion of subjects completing follow-up at 30 days post-procedure | 30 days post-procedure
  Proportion of subjects completing follow-up at 30 days post-procedure
Proportion of subjects completing follow-up at 6 months post-procedure | 6 months post-procedure
  Proportion of subjects completing follow-up at 6 months post-procedure
Absolute change in vegetation size pre-procedure to post-procedure | Periprocedural/immediately post-procedure
  Absolute change in vegetation size immediately pre-procedure to immediately post-procedure, measured by comparing imaging performed immediately pre-procedure to imaging performed immediately post-procedure (TEE)
Percent change in vegetation size pre-procedure to post-procedure | Periprocedural/immediately post-procedure
  Percent change in vegetation size immediately pre-procedure to immediately post-procedure, measured by comparing imaging performed immediately pre-procedure to imaging performed immediately post-procedure (TEE)
Intraoperative survival | Periprocedural/immediately post-procedure
  Proportion of patients who survive the index procedure
In-hospital survival | Through hospital discharge, up to 6 months post-procedure
  Proportion of patients who survive to be discharged from the hospital
30-day survival | 30 days post-procedure
  30-day survival
6-month survival | 6 months post-procedure
  6-month survival
Absence of persistent bacteremia within 7 days post-procedure | 7 days post-procedure
  Absence of persistent bacteremia within 7 days post-procedure
Absence of persistent bacteremia within 30 days post-procedure | 30 days post-procedure
  Absence of persistent bacteremia within 30 days post-procedure
Absence of further right-sided valve intervention through 30 days post-procedure | 30 days post-procedure
  Absence of further right-sided valve intervention through 30 days post-procedure
Absence of further right-sided valve intervention through 6 months post-procedure | 6 months post-procedure
  Absence of further right-sided valve intervention through 6 months post-procedure
Increase in valvular regurgitation post-procedure | Periprocedural/immediately post-procedure
  Increase in valvular regurgitation (i.e., mild to moderate or severe; moderate to severe) measured on imaging performed immediately pre-procedure to imaging performed immediately post-procedure (TEE)
Increase in valvular regurgitation 7 days post-procedure | 7 days post-procedure
  Increase in valvular regurgitation 7 days post-procedure (TTE)
Increase in valvular regurgitation 30 days post-procedure | 30 days post-procedure
  Increase in valvular regurgitation 30 days post-procedure (TTE)
Increase in valvular regurgitation 6 months post-procedure | 6 months post-procedure
  Increase in valvular regurgitation 6 months post-procedure (TTE)
Hospital length of stay | Through hospital discharge, from date admitted to the hospital to date discharged from the hospital, up to 6 months post-procedure
  Number of days patients are in the hospital, from date admitted to date discharged from the hospital
Intensive Care Unit (ICU) length of stay | Through ICU discharge, from date admitted to the ICU to date discharged from the ICU, up to 6 months post-procedure
  Number of days patients are in the Intensive Care Unit (ICU), from date admitted to the ICU to date discharged from the ICU
Blood loss | Periprocedural/immediately post-procedure
  Amount of blood lost during the procedure (cc) per Investigator estimate
Transfusion secondary to periprocedural and post-procedural bleeding complications | Through hospital discharge, up to 6 months post-procedure
  Number of transfusions required secondary to periprocedural and post-procedural bleeding complications
Rate of Device-Related Adverse Events (AEs) | Through 6 months post-procedure
  The number and proportion of subjects who experienced at least one device-related adverse event during the study
All-cause mortality | Through 6 months post-procedure
  All-cause mortality
Rate of Major Bleeding | Through 6 months post-procedure
  The number and proportion of subjects who experienced at Major Bleeding
Rate of device- or procedure-related individual Adverse Events of Special Interest (AESI) | Through 6 months post-procedure
  AESI include: cardiac perforation, vascular perforation, dissection, pericardial effusion, cardiac tamponade, pulmonary embolism, arterial thrombosis, venous thrombosis, acute kidney injury, acute liver injury, microangiopathy, micro-thrombotic disease, systemic inflammatory response syndrome (SIRS), and hemolysis
Change in blood quality parameters | Through 30 days post-procedure
  Absolute difference and percent difference in blood quality parameters from baseline to post-procedure (immediately post-procedure), 7 days, hospital discharge, and 30 days